CLINICAL TRIAL: NCT07035730
Title: Post-stroke Gait Rehabilitation With a Unilateral Hip Exoskeleton: Clinical and Neuromuscular Outcomes
Brief Title: Post-stroke Gait Rehabilitation Using the SHAJA-R Exoskeleton
Acronym: SHAJA-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmelo Chisari (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other); Centro Riabilitativo Villa Beretta (Unknown); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor-Investigator, Carmelo Chisari, Associate Professor, University of Pisa
Organization: University of Pisa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0003812/2025
Record Dates: First submitted 2025-06-03; First posted 2025-06-25 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHAJA first, then conventional (Experimental): Patients will perform the SHAJA-assisted gait training during the first period of the trial followed by a conventional gait training during the second period of the trial
  Interventions: Device: Unilateral hip exoskeleton; Behavioral: Conventional gait training
- Conventional first, then SHAJA (Experimental): Patients will perform the conventional gait training during the first period of the trial followed by a SHAJA-assisted gait training during the second period of the trial
  Interventions: Device: Unilateral hip exoskeleton; Behavioral: Conventional gait training

INTERVENTIONS:
Device: Unilateral hip exoskeleton — Unilateral hip exoskeleton assisted gait training. Gait training will consist of overground walking with the exoskeleton SHAJA for 30-40 minutes.
Behavioral: Conventional gait training — Conventional gait training will consist of overground walking without the exoskeleton SHAJA for 30-40 minutes.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, reliability, and short-term effectiveness of SHAJA-based training in improving walking velocity and endurance in post-stroke patients.

The main questions it aims to answer are:

* Does the SHAJA-based training improve walking velocity and endurance in post-stroke patients compared to conventional gait training?
* Is the SHAJA exoskeleton safe and reliable?

Researchers will compare the SHAJA-based training to a conventional gait training to see if the former works to improve walking ability.

Participants will:

* Perform six SHAJA-assisted gait training sessions or six conventional gait training sessions
* Perform five assessment sessions

ELIGIBILITY:
Inclusion Criteria:

* cerebral stroke, at least 3 months from cerebral event
* ability to ambulate with no more than minimal contact assistance, even with aids (Functional Ambulation Classification, FAC >= 43)
* self-selected walking velocity in the range [0.3-0.85] m/s
* anthropometry consistent with the specifications of the tested devices
* gait impairments that may benefit from hip assistance, e.g. hip weakness in flexion and/or extension (Medical Research Council, MRC, Scale for Muscle Strength >2 and <5 for flexion and extension)

Exclusion Criteria:

* Modified Ashworth Scale >3 at the hip and/or ankle joints
* Poor cognitive skills (corrected Mini-Mental State Examination, MMSE < 21)
* inability to follow verbal 3 step commands
* severe aphasia causing inability to communicate with the investigators
* serious medical conditions (recent myocardial infarction in less than 3 months, uncontrolled congestive heart failure (CHF), uncontrolled hypertension, uncontrolled seizures)
* leg deep vein thrombosis less than 6 weeks ago
* other pre-existing neurological disorders (Parkinson's disease, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Dementia)
* severe anxiety or depression (State-Trait Anxiety Inventory-Y, STAI-Y > 44, and the Beck Depression Inventory-II, BDI-II > 19)
* severe osteoporosis
* severe hip / knee osteoarthritis with limitation of movement or significant pain
* use of a colostomy bag
* skin wounds, infection, or problems at device contact locations
* major orthopaedic surgery or fractures within the last 90 days (hip, knee, ankle, foot, spine)
* cardiac surgery within the last 3 months
* patient has recently or is currently participating in research that may influence, in PI's opinion, responses to study intervention
* pregnancy
* implanted cardiac devices, such as pacemakers or automatic defibrillators (AICD)
* use of assistive device that, in the PI's opinion, could interfere with SHAJA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of device-related adverse events | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1
Documenting device hardware and software malfunctions | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1
Changes in self-selected walking velocity (m/s) pre vs post Conventional training and SHAJA-assisted training interventions assessed with the 10 Metre Walk Test | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
Changes in fast walking velocity (m/s) pre vs post Conventional training and SHAJA-assisted training interventions assessed with the 10 Metre Walk Test | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
Changes in the difference between self-selected and fast walking velocity (delta m/s) pre vs post Conventional training and SHAJA-assisted training interventions assessed with the 10 Metre Walk Test | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
Changes in walking endurance (in minutes) pre vs post Conventional training and SHAJA-assisted training interventions assessed with a Walk Test | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1

SECONDARY OUTCOMES:
Changes in gait kinematics/kinetics pre vs post Conventional training and SHAJA-assisted training interventions assessed with a motion capture system | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
Changes in the execution time of the Timed-Up-and-Go (TUG) test pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
Changes in Berg Balance Scale pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
  The Berg Balance Scale ranges from 0 to 56, with higher scores indicating better performance
Changes in Motricity Index for Lower Limb pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
  The Motricity Index ranges from 0 to 100, with higher scores indicating better performance
Changes in Modified Ashworth Scale (MAS) pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
  The Modified Ashworth Scale ranges from 0 to 4, with lower scores indicating better outcome
Changes in Functional Ambulation Classification (FAC) pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the follow up, about 14 weeks after T1
  The Functional Ambulation Classification ranges from 1 to 6, with higher scores indicating better performance

OTHER OUTCOMES:
Changes in lower-limb muscle activity through superficial Electromyography (sEMG) pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1
Changes in lower-limb muscle synergies pre vs post Conventional training and SHAJA-assisted training interventions assessed by electromyography during walking | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1
Changes in cortico-cortical connectivity through superficial Electroencephalography (sEEG) pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1
Changes in cortico-muscular connectivity through sEMG and sEEG pre vs post Conventional training and SHAJA-assisted training interventions | From the pre-training evaluation (T1) to the second post-training evaluation, about 3 months after T1

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro Riabilitativo Villa Beretta, Costa Masnaga, Italy
  - SD Neuroriabilitazione - Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication